CLINICAL TRIAL: NCT04849130
Title: DynMPFL - Comparison of Dynamic and Static Medial Patellofemoral Ligament Operation Technique for Recurrent Patellar Dislocation
Brief Title: Comparison of Dynamic and Static Medial Patellofemoral Ligament Operation Technique for Recurrent Patellar Dislocation
Acronym: DynMPFL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2020-02701; mu21Egloff
Record Dates: First submitted 2021-04-07; First posted 2021-04-19 (Actual); Last update posted 2025-04-22 (Actual); Status verified 2025-04

CONDITIONS: Patellar Instability
Keywords: chronic patellar instability; static medial patellofemoral ligament (MPFL) reconstruction; static reconstruction technique according to Schöttle; dynamic medial patellofemoral ligament (MPFL) reconstruction; patellofemoral ligament reconstruction; patella dislocation; Patella-Instability-Severity (PIS) score; dynamic reconstruction technique according to Becher
MeSH Terms: conditions — Patellar Dislocation

STUDY DESIGN:
Intervention Model Description: Multicentre prospective longitudinal randomized clinical trial
Who Masked: Participant, Outcomes Assessor
Masking Description: Study assessments blinded by separating the clinicians performing the surgery and independent blind observers assessing the study data. Patients will be blinded to the surgery procedure.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Static reconstruction technique according to Schöttle (Active Comparator): Static reconstruction technique according to Schöttle
  Interventions: Procedure: Static reconstruction technique according to Schöttle
- Dynamic reconstruction technique according to Becher (Active Comparator): Dynamic reconstruction technique according to Becher
  Interventions: Procedure: Dynamic reconstruction technique according to Becher

INTERVENTIONS:
Procedure: Static reconstruction technique according to Schöttle — In static MPFL reconstruction, a graft (harvested autologous gracilis tendon or allogen transplant) is attached to the femoral and patellar bones using tunnels, screws, and/or anchors.
  Arms: Static reconstruction technique according to Schöttle
Procedure: Dynamic reconstruction technique according to Becher — Dynamic MPFL procedure by detaching and reinserting only the distal part of a hamstring muscle to the patella and leaving the proximal tendon attached to its muscle. This way the patella position can be adjusted dynamically by hamstring contraction.
  Arms: Dynamic reconstruction technique according to Becher

SUMMARY:
This study is to evaluate whether the dynamic Medial Patellofemoral Ligament (MPFL) reconstruction as described by Becher is a successful operation technique to prevent patella instability and restore quality of life. It is to assess and compare clinical and functional outcomes of dynamic and static medial patellofemoral ligament reconstruction

DETAILED DESCRIPTION:
The recurrent dislocation rate of conservatively treated chronic patellar instability is high, therefore, it is recommended to manage it surgically. A frequently used surgical technique is static medial patellofemoral ligament (MPFL) reconstruction (e.g. Schöttle-technique). A novel dynamic surgical technique according to Becher was developed, addressing the most common complications occurring in static reconstruction, which are malpositioning and overtensioning of the graft. This study is to assess and compare clinical and functional outcomes of dynamic and static medial patellofemoral ligament reconstruction.

ELIGIBILITY:
Inclusion Criteria:

* Patients treated with isolated dynamic (operation procedure according to Becher et al.using the gracilis tendon) or static MPFL plastic (operation procedure according to Schöttle et al. using the gracilis tendon). MPFL reconstruction will be performed in patients with preceding patella dislocation with: 1) a Patella-Instability-Severity (PIS) score ≤ 3 with concomitant flake fracture or 2) a PIS score ≥ 4 with clinical asymptomatic trochlea dysplasia (patella stability between 30°-60° knee flexion) without other clinically relevant static risk factors.
* Closed growth plates

Exclusion Criteria:

* Combined procedures with trochleoplasty (high grade trochlea dysplasia, type Dejour C,D with clinical instability between 30° and 60° of knee flexion)
* combined procedures with cartilage transplantation
* High grade patellofemoral arthritis (Kellgren Lawrence score ≥3)
* combined procedures with femoral or tibial osteotomy
* Clinically eminent valgus axis (>15° valgus)
* Femoral internal rotation >20°, tibial external rotation >40°
* Instability of the cruciate or collateral ligaments
* Known significant musculoskeletal disease
* Cognitive impairment

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-05-10 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Change in Kujala score | up to 24 months
  Patient reported knee function and anterior knee pain as assessed with the Kujala score at preoperative screening, at the hospitalization time and four postoperative follow ups . The Kujala scale consists of 13 questions covering a range of physical symptoms and limitations that are presented in a multiple choice answer format, with a different point value assigned to each answer. The maximum score is 100, with higher scores indicating better function.

SECONDARY OUTCOMES:
Number of recurrent patella dislocation | From MPFL surgery to occurring recurrent patella dislocation (up to 24 months)
  Surgical outcome: recurrent patella dislocation.
Number of revision surgery | From MPFL surgery to occurring revision surgery (up to 24 months)
  Surgical outcome: revision surgery.
Number of complications (other than revision surgery, e.g. infection, wound healing disorder) | From MPFL surgery to occurring complication (up to 24 months)
  Surgical outcome: complications (other than revision surgery, e.g. infection, wound healing disorder).
Change in Banff-II-score from preoperative screening, at the hospitalization time and four postoperative follow ups | up to 24 months
  The Banff Patella Instability Instrument (BPII) is a disease-specific health-related quality of life score. It is a patient-reported, disease-specific QOL score that consists of 23 questions across five domains covering symptoms/physical complains, work-related concerns, recreational activity and sport participation/competition, lifestyle, and social/emotional. Patients mark their answers on a visual analogue scale measuring 100 mm in length. Each item is equally weighted with the final score calculated as an average of the scores from all answered items. A higher score reflects a higher QOL.
Change in International Knee Documentation Committee (IKDC)-2000 from preoperative screening, at the hospitalization time and four postoperative follow ups | up to 24 months
  The IKDC includes 18 questions covering three domains: symptoms, physical activity, and function. The items are answered on Likert scales of varying values. IKDC scores are calculated by dividing the total score by the highest possible score for the items answered, and multiplying by 100, with higher scores indicating better function.
Change in EQ-5D-5L from preoperative screening, at the hospitalization time and four postoperative follow ups EQ-5D- EQ-5D-5L | up to 24 months
  The EQ-5D descriptive system comprises five dimensions: mobility, self-care, usual activities, pain and discomfort, and anxiety and depression. The five levels in each dimension are worded as (1) 'not /no problems', (2) 'slight problems', (3) 'moderate problems', (4) 'severe problems', and (5) 'unable to' (mobility, self-care, usual activities), 'extreme' (pain/depression), or 'extremely' (anxiety/depression).
Change in pain level using the numeric rating scale from preoperative screening, at the hospitalization time and four postoperative follow ups | up to 24 months
  It is usually presented as a 100-mm horizontal line on which the patient's pain intensity is represented by a point between the extremes of "no pain at all" and "worst pain imaginable."
Operation time | During MPFL surgery (up to 1 day)
  Operation time
Hospitalization time | During hospitalization (up to 1 month)
  Length of hospital stay Length of hospital stay
Change in gait asymmetry | Preoperatively and 1 year postoperative
  Instrumented gait analysis (by EMG) on a treadmill with an embedded plantar pressure plate and on an overground walkway with two embedded force plates.
Change in isokinetic muscle strength | Preoperatively and 1 year postoperative
  Muscle strength will be measured bilaterally using a dynamometer.
Change in timing of muscle activity | Preoperatively and 1 year postoperative
  Timing of the gracilis muscle will be assessed as on- and offset relative to the gait cycle. Gracilis onset will be determined as the time when the processed EMG signal exceeded a threshold of three standard deviations above a baseline mean and as offset, when the processed EMG signal falls below a threshold of three standard deviations above a baseline mean.
Change in single legged drop test | Preoperatively and 1 year postoperative
  Standing erect upon only the tested leg with the foot in neutral position, participants will step off a 30 cm high platform placed 11 cm from the edge of the force-plate. Participants will be instructed to land in the centre of the force-plate on the tested leg only.

CONTACTS AND LOCATIONS:
Overall Officials: Christian Egloff, PD Dr. med., Principal Investigator — Department of Orthopaedics and Traumatology, University Hospital Basel
Locations (2):
- Switzerland (2):
  - Department of Orthopaedics and Traumatology, University Hospital Basel, Basel
  - Department of Orthopaedics and Traumatology, Swiss Altius Medical Clinic, Rheinfelden

REFERENCES:
- [Derived] Bartsch A, Nuesch C, Rieger B, Mundermann A, Egloff C. Dynamic versus static medial patellofemoral ligament reconstruction technique in the treatment of recurrent patellar dislocation: a randomized clinical trial protocol. J Orthop Surg Res. 2022 Jul 10;17(1):345. doi: 10.1186/s13018-022-03158-6. PMID 35818060